CLINICAL TRIAL: NCT05221632
Title: Accelerated cTBS and 1HZ-rTMS in the Treatment of Obsessive-compulsive Disorder With Individualized Stimulation Target
Brief Title: Accelerated Continue Theta-burst Stimulation (acTBS)Treatment for Obsessive Compulsive Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Zhu, A/Prof., Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: precise high-dose OCD
Record Dates: First submitted 2022-01-03; First posted 2022-02-03 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Obsessive-Compulsive Disorder; Accelerated Continue Theta-burst Stimulation; Transcranial Magnetic Stimulation; Functional Magnetic Resonance Imaging
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- accelerated continue theta-burst stimulation (Experimental): Fifty intermittent TBS sessions (1800 pulses per session, 50 minute inter-session interval ) were delivered as ten daily sessions over five consecutive days at 80% resting motor threshold (RMT). The MRI data set should be collected before the first cTBS session and after the last cTBS session.
  Interventions: Device: Accelerated transcranial magnetic stimulation with real coil
- 1-HZ repetition transcranial magnetic stimulation Stimulation (Active Comparator): The repetition transcranial magnetic stimulation(rTMS) lasted 30 mins and delivered at 1 Hz with 1s duration, a total of 1800 pulses at 80% of the rest motor threshold (RMT) . MRI dataset should be acquired before the first rTMS session and after the last rTMS session.
  Interventions: Device: Transcranial magnetic stimulation with real coil
- accelerated continue theta-burst stimulation (sham) (Sham Comparator): Fifty intermittent TBS sessions (1800 pulses per session, 50 minute inter-session interval ) were delivered as ten daily sessions over five consecutive days at 80% resting motor threshold (RMT). The MRI data set should be collected before the first cTBS session and after the last rTMS session. No actual magnetic stimulation was applied on the head of the volunteers. MRI dataset should be acquired before the first cTBS session and after the last cTBS session.
  Interventions: Device: Transcranial magnetic stimulation with sham coil

INTERVENTIONS:
Device: Accelerated transcranial magnetic stimulation with real coil — The stimulation mode of TMS is accelerated continue theta-burst stimulation.
  Arms: accelerated continue theta-burst stimulation
Device: Transcranial magnetic stimulation with real coil — The stimulation mode of TMS is 1-Hz repetitive Transcranial magnetic stimulation .
  Arms: 1-HZ repetition transcranial magnetic stimulation Stimulation
Device: Transcranial magnetic stimulation with sham coil — The stimulation mode of TMS is accelerated continue theta-burst stimulation, but without active stimulation.
  Arms: accelerated continue theta-burst stimulation (sham)

SUMMARY:
The therapeutic effects of high-dose accelerated continue theta-burst stimulation (acTBS) and 1-Hz repetitive transcranial magnetic stimulation (rTMS) on obsessive-compulsive disorder (OCD) and its neural mechanism were investigated by functional MRI.

DETAILED DESCRIPTION:
All patients underwent a medical evaluation that included physical examination and routine laboratory studies before and after transcranial magnetic stimulation (rTMS) treatment. Patients were randomly allocated to 1-Hz rTMS group，acTBS group and sham group. Patients ware allocated by random number. The decision to enroll a patient was always made prior to randomization. The 1-Hz rTMS group received one round of stimulation every day for 30 minutes with a total stimulation of 1800 pulses for 5 consecutive days. Patients in the acTBS group received 10 two-minute rounds of stimulation each day, spaced 50 minutes apart, with a total of 18,000 pulses for five days.

Before the TMS treatment, Y-BOCS, Obsessions Symptom Scale revised (OCI-R), Hamilton Depression Scale (HAMD-17) and Hamilton Anxiety Scale (HAMA-14) were obtained by a trained investigator to assess baseline severity and other symptoms. The patients had receiving a battery measure of neuropsychological tests (standardized tests to investigate their cognitive problems, anxiety and depressive symptoms in daily life), magnetic resonance imaging scan in multimodalities。

After the last treatment, Yale-Brown Obsessive-Compulsive Scale (Y-BOCS), OCI-R, HAMD-17 and HAMA-14 were obtained, as well as the Global Index of Safety to assess adverse events of the treatment. Patients were instructed to focus their answers on the past 5 days.The patients had also receiving a battery measure of neuropsychological tests and magnetic resonance imaging scan in multimodalities.

Participants were interviewed for two and four weeks after their last treatment to obtain a Y-BOCS score, and they were asked to focus their answers on the past week.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obsessive-compulsive disorder
* Voluntarily participated and cooperated with the experiment.

Exclusion Criteria:

* History of significant head trauma or neurological disorders.
* Alcohol or drug abuse.
* Organic brain defects on T1 or T2 images.
* History of seizures or unexplained loss of consciousness.
* Family history of medication refractory epilepsy.
* Recent aggression or other forms of behavioral dyscontrol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-01-06 (Actual); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptom improvement assessed by the Yale-Brown Obsessive Compulsive Scale | pre-treatment; 1 day post-treatment; Change from baseline score at 1 month
  The Yale-Brown Obsessive Compulsive Scale is a test to rate the severity of obsessive-compulsive disorder symptoms, which measures obsessions separately from compulsions. The scale includes 10 items, the first 5 items are evaluated obsessions, the rest are assessments compulsions. Each item 0-4 points, a total of 40 points. The lower the score, the better the outcome.

SECONDARY OUTCOMES:
Obsessive Compulsive Inventory-Revised (OCI-R) | pre-treatment; 1 day post-treatment
  a simplified version of the OCI for self-assessment of Obsessive symptoms, Revised to include only 18 items from 42 items in the original Obsessive Compulsive Questionnaire. Divided into six obsessional subscales, respectively washing (5, 11, 17), obsessional thinking (6, 12, 18), storage (1, 7, 13), sorting (3, 9, 15), check (2, 8, 14), mixed (4, 10, 16), can be very good to distinguish the characteristics of different obsessional symptoms. Each item was assessed on a five-point scale of 0 to 4, with 0 being "not at all" and 5 being "extremely painful," and participants were asked to tick a number that best described the extent of their pain or distress on a scale of 0 to 72, with higher scores indicating more severe obsessive-compulsive symptoms. The questionnaire is simple and easy to understand. It can objectively evaluate individual obsessive-compulsive symptoms from six dimensions, with high reliability (0.82) and validity (0.81).
Hamilton Depression Scale（HAMD） | pre-treatment; 1 day post-treatment
  Hamilton Depression Scale（HAMD）: An assessment of depressive mood status with 17 questions on a Scale of 0 to 4.
Hamilton Anxiety Scale（HAMA） | pre-treatment; 1 day post-treatment
  Hamilton Anxiety Scale（HAMA）：a scale of 14 questions on a scale of 0 to 4 on a 5 scale.
Stroop word test | pre-treatment; 1 day post-treatment
  To measure the conflict suppression ability of the subjects, consisting of three groups of cards, namely dot, word and color word. The subjects were asked to read the color as quickly and accurately as possible, and record the response time and accuracy. Behavioral indicators :(Stroop interference effects, SIE)= reaction time of color word - reaction time of word.
Behavioral index TMT=TMT-B reaction time - TMT-A reaction time. | pre-treatment; 1 day post-treatment
  Evaluate the executive function of the subjects, including attention, memory, thinking flexibility, reasoning, conversion and other broad executive function components, including A and B. TMT is simple and involves less cognitive involvement. TMT-B involves response inhibition and attentional switching. The task required the subjects to complete the connection according to certain rules and record the reaction time. Behavioral index TMT=TMT-B reaction time - TMT-A reaction time.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

REFERENCES:
- [Derived] Jiang J, Wan K, Liu Y, Tang Y, Tang W, Liu J, Ma J, Xue C, Chen L, Qian H, Liu D, Shen X, Fan R, Wang Y, Wang K, Ji G, Zhu C. A Controlled Clinical Study of Accelerated High-Dose Theta Burst Stimulation in Patients with Obsessive-Compulsive Disorder. Neural Plast. 2023 Dec 7;2023:2741287. doi: 10.1155/2023/2741287. eCollection 2023. PMID 38099081